CLINICAL TRIAL: NCT05373433
Title: A Randomized, Double-blind, Placebo-controlled, Phase II/III Clinical Study Evaluating the Efficacy and Safety of SSD8432 in Combination With Ritonavir in Adult Subjects With Mild/Common COVID-19
Brief Title: To Evaluate SSD8432/Ritonavir in Adults With COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B02B11101-302
Record Dates: First submitted 2022-05-12; First posted 2022-05-13 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SIM0417; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): SSD8432 750mg and Ritonavir 100mg
  Interventions: Drug: SSD8432 750mg
- Control group (Placebo Comparator): SSD8432 placebo and Ritonavir placebo
  Interventions: Drug: SSD8432 placebo

INTERVENTIONS:
Drug: SSD8432 750mg — Experimental group:SSD8432 750mg and Ritonavir 100mg, Day1--Day5,BID
  Other Names: Ritonavir 100mg
  Arms: Experimental group
Drug: SSD8432 placebo — Control group :SSD8432 placebo and Ritonavir placebo, Day1--Day5,BID
  Other Names: Ritonavir placebo
  Arms: Control group

SUMMARY:
This is a randomized, double-blind, placebo-controlled, phase II/III clinical study to evaluate the efficacy and safety of SSD8432 in combination with ritonavir in adult subjects with mild/common COVID-19.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, phase II/III clinical study to evaluate the efficacy and safety of SSD8432 in combination with ritonavir in adult subjects with mild/common COVID-19.

This study plan to enroll 670 mild or common type adult COVID-19 subjects, Randomly assigned to the experimental group and the control group according to 1:1, experimental group:335subjects will receive SSD8432 and Ritonavir; control group :335subjects will receive SSD8432 placebo and Ritonavir placebo.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 and ≤80 years old, male or female.
2. Initial positive test of SARS-CoV-2 within 5 days of randomization.
3. mild or common type of COVID-19.
4. Initial onset of COVID-19 signs/symptoms within 3 days of randomization.
5. Fever or 1 respiratory symptom of COVID-19 on random day
6. Subjects without high risk factors
7. Subjects with at least one high-risk factor

Exclusion Criteria:

1. Transnasal high-flow oxygen therapy or non-invasive ventilation, invasive mechanical ventilation, or ECMO is required or anticipated to be urgently required.
2. Prior to current disease episode, any confirmed SARS-CoV-2 infection.
3. Known medical history of active liver disease (other than nonalcoholic hepatic steatosis).
4. Receiving dialysis or have known moderate to severe renal impairment.
5. Known human immunodeficiency virus (HIV) infection.
6. Suspected or confirmed concurrent active systemic infection other than COVID-19 that may interfere with the evaluation of response to the study intervention.
7. Oxygen saturation of ≤ 93% on room air obtained at rest within 24 hours prior to randomization..
8. Treatment with antivirals against SARS-CoV-2 within 14 days.
9. Current or expected use of any medications or substances that are highly dependent on CYP3A4 for clearance.
10. Concomitant use of any medications or substances that are strong inducers of CYP3A4 are prohibited within 28 days.
11. Has received or is expected to receive COVID-19 monoclonal antibody, convalescent COVID-19 plasma or other prohibited concomitant medication.
12. Females who are pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2022-05-26 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Viral load | Baseline through Day6
  Change from baseline in viral load of SARS-CoV-2 in throat swabs by RT-PCR on Day 6 (after last dose)
Time to Sustained Alleviation | Baseline through Day28
  Time to Sustained Alleviation of 5 COVID-19 signs/symptoms

SECONDARY OUTCOMES:
Viral load | Baseline through Day28
  Changes of viral load compared to the baseline
Time to Sustained Alleviation | Baseline through Day28
  Time to Sustained Alleviation of target COVID-19 signs/symptoms
Proportion of participants progress to a worsening status(higher score) | Baseline through Day28
  WHO clinical progress scale(0 to 10)
Adverse events | Baseline through Day28
  Frequency of TEAE
Maximum plasma concentration(Cmax) | Baseline through Day5
  Plasma concentration of SSD8432

CONTACTS AND LOCATIONS:
Overall Officials: Yumei Yang, Doctor, Study Director — Jiangsu Xiansheng Pharmaceutical Co.,

IPD SHARING:
Plan to Share IPD: No